CLINICAL TRIAL: NCT04169347
Title: Phase II Pilot Study of FOLFOXIRI Plus Panitumumab in Metastatic RAS Wild-type, Left-sided Colorectal Cancer
Brief Title: FOLFOXIRI Plus Panitumumab in Metastatic RAS Wild-type, Left-sided Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Criterium, Inc. (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Panit7156
Record Dates: First submitted 2019-09-24; First posted 2019-11-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer Metastatic
MeSH Terms: interventions — Oxaliplatin; Irinotecan; Leucovorin; Panitumumab

STUDY DESIGN:
Intervention Model Description: Multicenter open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (Other): This is an open label study single arm
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Oxaliplatin — 2 week cycles
  Other Names: Irinotecan; Leucovorin; Panitumumab

SUMMARY:
This is a phase II, open-label, non-randomized study in subjects with histologically confirmed diagnosis of left-sided RAS WT advanced adenocarcinoma of the colon or rectum who have not received prior systemic therapy for metastatic disease.

DETAILED DESCRIPTION:
This trial is designed to evaluate the efficacy of the combination of FOLFOXIRI and panitumumab as first-line therapy in patients with metastatic, left-sided, RAS WT CRC. The research hypothesis is that in this cohort of patients, the combination of triplet chemotherapy and anti-EGFR therapy will confer higher response rates and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have signed an approved informed consent.
2. Histologically confirmed diagnosis of advanced adenocarcinoma of the colon or rectum.
3. No previous systemic chemotherapy for metastatic disease

   * Subjects who have had prior adjuvant chemotherapy for non-metastatic disease are eligible if more than six months have elapsed after completing therapy
   * Subjects treated with adjuvant chemotherapy who relapse within six months after completion will not be eligible.
4. Bidimensionally measurable disease as defined in Section 3.3.1.
5. RAS wild-type tested in

   * KRAS exon 2 (codons 12/13)
   * KRAS exon 3 (codons 59/61)
   * KRAS exon 4 (codons 117/146)
   * NRAS exon 2 (codons 12/13)
   * NRAS exon 3 (codons 59/61)
   * NRAS exon 4 (codons 117/146)
6. ECOG Performance Status 0-1 (Appendix 1).
7. Recovery in full, from any previous surgical procedure.
8. Subjects >=18 years of age. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 6 months after the study in such a manner that the risk of pregnancy is minimized.

   WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or is not postmenopausal.

   WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.
9. Creatinine clearance ≥ 50 ml/min or serum creatinine ≤ 1.5 x upper limit of normal.
10. Bilirubin ≤ 1.5 x upper limit of normal
11. AST, ALT ≤ 2.5 x upper limit of normal in absence of liver metastases, or ≤ 5 x upper limit of normal in presence of liver metastases,
12. Albumin within normal institutional limits
13. Magnesium ≥ lower limit of normal; calcium ≥ lower limit of normal .
14. Absolute Neutrophil Count > 1500/mm3 and platelets > 100,000/mm3.

Exclusion Criteria:

1. WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 6 months after the study. Subjects who are men must also agree to use effective contraception.
2. Women who are pregnant or breastfeeding.
3. Women with a positive pregnancy test on enrollment or prior to study drug administration.
4. Subjects with >grade 1 neuropathy except for loss of tendon reflex.
5. Any active or uncontrolled infection.
6. Clinically significant cardiovascular disease (myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 6 months before enrollment
7. Past or current history of malignancies except for the indication under this study and curatively treated:

   * Basal and squamous cell carcinoma of the skin
   * In-situ carcinoma of the cervix
   * Other malignant disease without recurrence after at least 3 years of follow-up
8. History or evidence upon physical examination of CNS disease unless adequately treated (e.g. primary brain tumor, seizure not controlled with standard medical therapy, brain metastases or history of stroke).
9. Clinically relevant interstitial lung disease (pneumonitis, pulmonary fibrosis, evidence of interstitial lung disease on baseline chest CT scan)
10. Allogeneic transplantation requiring immunosuppressive therapy.
11. Severe non-healing wounds, ulcers or bone fractures.
12. Evidence of bleeding diathesis or coagulopathy.
13. Patients not receiving therapeutic anticoagulation must have an INR < 1.5 x ULN and aPTT < 1.5 x ULN within 7 days prior to randomization. The use of full-dose anticoagulants is allowed as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose for anticoagulants for at least two weeks.
14. Concomitant therapy with certain anti-viral medicines (sorivudine and brivudine or analogue compounds).
15. Major surgical procedure, open biopsy, nor significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study except for surgery for colorectal cancer with curative intent and central venous line placement for chemotherapy administration.
16. Subjects with known allergy to the study drugs or to any of its metabolites.
17. Known DPD deficiency.
18. Current or recent (within the 28 days prior to starting study treatment) treatment of another investigational drug or participation in another investigational study.
19. Known grade III/IV allergic reaction against monoclonal antibodies.
20. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy/objective response rate | Through progression of disease, on average 6 months.
  Evaluate the efficacy/objective response rate of the combination of FOLFOXIRI and panitumumab as first-line therapy for metastatic left-sided, RAS WT CRC.

SECONDARY OUTCOMES:
Evaluating progression free survival (PFS) | Through progression of disease, on average 6 months.
  The secondary efficacy endpoints include time to progression and overall survival. Kaplan-Meier estimates will be calculated for time to progression and overall survival, and medians, along with two-sided 95% confidence intervals, will be reported.
Evaluating overall survival (OS) | Through progression of disease, on average 6 months.
  The secondary efficacy endpoints include time to progression and overall survival. Kaplan-Meier estimates will be calculated for time to progression and overall survival, and medians, along with two-sided 95% confidence intervals, will be reported.
Evaluating toxicity of this regimen | Through progression of disease, on average 6 months.
  Subjects will be evaluated for toxicity/safety profile using CTCAE v4
Evaluating radiographic tumor regression | Through progression of disease, on average 6 months.
  Subjects will be evaluated for response according to the tumor response measured with RECIST v1.1a
Evaluating for the velocity of tumor response to this regimen | Patients will be followed until death or 5 years
  Exploratory objectives include measuring circulating tumor DNA to assess for clinical response and velocity of response.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Hochster, MD, Principal Investigator — Lead Site PI
Locations (8):
- United States (8):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Yale Cancer Center, New Haven, Connecticut
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Kansas University Cancer Center, Westwood, Kansas
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Laura & Isaac Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Swedish Cancer Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No